CLINICAL TRIAL: NCT03726177
Title: Comparison of Two Doses (81 mg Versus 162mg) of Aspirin for the Prevention of Preeclampsia in High-Risk Pregnant Women: A Randomized Controlled Trial
Brief Title: Aspirin for Prevention of Preeclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu 194/7/18
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Preeclampsia
Keywords: preeclampsia; low dose aspirin; high risk pregnancy
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: This will be a randomized control trial to estimate the efficacy of two doses (80 mg versus 160 mg) of aspirin for prevention of preeclampsia in High-Risk Pregnant Women identified in the first trimester to be at high risk.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: both participants and researchers will be blinded to the intervention given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aspirin 162 mg (Active Comparator): Aspirin 81mg two tablet once a day from recruitment until 37 weeks or labor whichever comes first
  Interventions: Drug: aspirin 162 mg
- aspirin 81 mg plus placebo (Active Comparator): Aspirin 81mg two tablet once a day from recruitment until 37 weeks or labor whichever comes first plus placebo one tablet once a day from recruitment until 37 weeks or labor whichever comes first
  Interventions: Drug: aspirin 81 mg; Drug: placebo

INTERVENTIONS:
Drug: aspirin 162 mg — Aspirin 81mg two tablet once a day from recruitment until 37 weeks or labor whichever comes first
  Other Names: Active Comparator
  Arms: aspirin 162 mg
Drug: aspirin 81 mg — Aspirin 81mg one tablet once a day from recruitment until 37 weeks or labor whichever comes first
  Other Names: active comparator
  Arms: aspirin 81 mg plus placebo
Drug: placebo — placebo one tablet once a day from recruitment until 37 weeks or labor whichever comes first
  Other Names: Placebo to asprin
  Arms: aspirin 81 mg plus placebo

SUMMARY:
Prophylaxis with low-dose aspirin has been recommended to prevent preeclampsia, the rationale being that hypertension and abnormalities of coagulation in this disease are caused in part by an imbalance between vasodilating and vasoconstricting prostaglandins. Low-dose aspirin therapy inhibits thromboxane production more than prostacyclin production and therefore should protect against vasoconstriction and pathologic blood coagulation in the placenta. Initially, several single-center trials, mostly among women at increased risk for preeclampsia, demonstrated a substantial reduction in the risk of proteinuric hypertension as well as reductions in the incidences of preterm birth, infants small for gestational age, and perinatal death,

DETAILED DESCRIPTION:
This will be a randomized control trial to estimate the efficacy of two doses (80 mg versus 160 mg) of aspirin for prevention of preeclampsia in High-Risk Pregnant Women identified in the first trimester to be at high risk.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women presenting prior to 17+0 weeks' gestation.
* Moderate to high risk of preeclampsia.
* One or more of the following: previous history of preeclampsia, antiphospholipid antibodies, pre-existing diabetes, pre-existing hypertension, pre-existing renal disease, autoimmune disease, nulliparity, family history of preeclampsia, elevated BMI > 25, and maternal age <20 or >35.
* Give written informed consent.

Exclusion Criteria:

* Multiple gestations,
* fetal aneuploidy
* major fetal structural anomaly
* bleeding disorder
* allergy to aspirin
* women already on aspirin or heparin.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The population of interest involves women attending the study hospital for antenatal care and delivery
Enrollment: 600 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With early Preeclampsia | 6 months
  The number of cases of preeclampsia that appear in both groups before 34 weeks of pregnancy.Blood pressure greater than 140/90 on 2 occasions 6 hrs apart and significant proteinuria (greater than 300 mg in 24 hrs) before 34 weeks gestation

SECONDARY OUTCOMES:
Prevention of preeclampsia between 37 and 41 | 6 months
  The number of cases of preeclampsia that appear in both groups between 37 and 41 weeks of pregnancy.
The number of cases of Fetal Growth Restriction | 6 months
  The number of cases of fetal growth restriction, defined as a fetal weight below the 10th percentile and an abnormal umbilical cord doppler that appear in both groups at any given time during pregnancy.
The number of cases of preterm birth | 6 months
  The number of cases delivered before 37 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No